CLINICAL TRIAL: NCT06354218
Title: A Single Arm, Prospective, Exploratory, Single Center Phase II Clinical Study of Serplulimab Combined With Synchronous Radiochemotherapy for the Treatment of Locally Advanced Esophageal Squamous Cell Cancer in Elderly Patients With Non Surgical Resectable Lesions Research Plan
Brief Title: Serplulimab Combined With Concurrent Chemoradiotherapy for Locally Advanced Treatment Esophageal Cancer in Old Age
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GXL-005
Record Dates: First submitted 2024-04-03; First posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Esophageal Carcinoma
Keywords: Serplulimab; Concurrent chemoradiotherapy
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Assigned Interventions (Experimental): Treatment options Serplulimab （4.5mg/Kg every 3 weeks）combined with chemoradiotherapy (Oral chemotherapy with the tigio regimen is given on days 1 to 2 of radiotherapy, with the drug dose 40-60mg BID, and the oral tigio course from Monday to Friday is synchronized with radiation therapy) for the treatment of locally advanced elderly esophageal cancer patients, in which the tigio regimen with good clinical tolerability was selected for chemotherapy to evaluate the short-term efficacy and toxic side effects
  Interventions: Drug: Serplulimab

INTERVENTIONS:
Drug: Serplulimab — Serplulimab （4.5mg/Kg every 3 weeks）
  Other Names: HLX-10LX

SUMMARY:
This study is a Single Arm, Prospective, Exploratory, Single Center Phase II Clinical Study to evaluate the effectiveness of the combination of Serplulimab and Concurrent Chemoradiotherapy in the treatment of elderly patients with locally advanced esophageal cancer who cannot be treated surgically.Subjects can be enrolled into this study only if they meet inclusion criteria and do not meet exclusion criteria.

DETAILED DESCRIPTION:
It is expected that 50 patients will be enrolled, and patients who meet the enrollment criteria will undergo esophagoscopy, esophageal barium meal examination, chest contrast-enhanced CT, abdominal ultrasound, electrocardiogram, blood routine, whole body bone scan, liver and kidney function and other examinations before treatment, and esophageal ultrasound if necessary. Patients who received esophageal ultrasound were staged by esophageal ultrasound results, and those without esophageal ultrasound were mainly staged according to the cervical chest and epigastric contrast CT and esophageal barium plates, and clinical staging was performed according to the AJCC staging standard. After the combination of Serplulimab and concurrent chemoradiotherapy, adverse reactions and efficacy evaluation were observed. The expected result is that the local control rate of Serplulimab combined with chemoradiotherapy is improved in patients with locally advanced elderly esophageal squamous cell carcinoma, and there is no significant increase in adverse reactions, and serological indicators such as PDL-1 CPS can be used as prognostic indicators for esophageal malignancy and have certain guiding significance for treatment. PD-1 monoclonal antibody can be used in locally advanced elderly esophageal cancer patients who cannot tolerate chemotherapy, with good short-term efficacy and tolerable toxic side effects, which further provides reference value for clinical guidance.

ELIGIBILITY:
Inclusion Criteria:

* 1. The patient voluntarily participated in this study, signed an informed consent form, had good compliance, and cooperated with follow-up; 2. Age 75 and above, both male and female; 3. Patients with locally advanced esophageal squamous cell carcinoma confirmed by histology and clinically classified as stage II-IVa that cannot be surgically removed (including non resectable, contraindications to surgery, or refusal to undergo surgery) (according to the 8th edition of AJCC staging, the pre-treatment clinical staging is cT1N2-3M0, cT2-4bN0-3M0); 4. PDL1 detection result CPS ≥ 1 5. There are measurable and/or unmeasurable lesions that meet the criteria for evaluating the efficacy of solid tumors (RECIST 1.1); 6. Have not received any systematic anti-tumor treatment in the past (including but not limited to systemic chemotherapy, radiotherapy, molecular targeted drug therapy, immunotherapy, biological therapy, local treatment, and other research treatment drugs); 7. ECOG: 0-1 points (see Attachment 1); 8. It is recommended to provide fresh or archived tumor tissue samples within 6 months (fresh samples are preferred) for biomarker analysis (such as PD-L1). The sample type is a formalin fixed, paraffin embedded [FFPE] tumor tissue block or at least 5 unstained, 3-5 thick pieces μ FFPE tumor tissue slice of m; 9. Expected survival time ≥ 3 months; 10. The functions of important organs meet the following requirements (no blood components or cell growth factors are allowed to be used 2 weeks before the start of screening examination): Absolute neutrophil count (ANC) ≥ 1.5 × 109/L; Platelets ≥ 100 × 109/L; Hemoglobin ≥ 9g/dL; Serum albumin ≥ 2.8g/dL; Total bilirubin ≤ 1.5 x ULN, ALT, AST, and/or AKP ≤ 2.5 x ULN; Serum creatinine ≤ 1.5 × ULN or creatinine clearance rate ≥ 60mL/min (calculated according to Cockcroft Gault formula, see Annex 2); International standardized ratio (INR) and activated partial thromboplastin time (APTT) ≤ 1.5 × ULN (for stable dose anticoagulant therapy such as low molecular weight heparin or warfarin, and INR can be screened within the expected therapeutic range of anticoagulants);

Exclusion Criteria:

* 1. History of esophageal cancer surgery; 2. Previous history of fistula caused by primary tumor infiltration; 3. There is a higher risk of gastrointestinal bleeding, esophageal fistula, or esophageal perforation; 4. Subjects with poor nutritional status and a weight loss of ≥ 10% within the first two months of screening showed no significant improvement after management and intervention; 5. Has undergone major surgery or had serious trauma within the first 4 weeks prior to the use of the investigational drug; 6. There are uncontrollable pleural effusion, pericardial effusion, or ascites that require repeated drainage; 7. Have received or are currently receiving any of the following treatments in the past:

  1. Anti PD-1 or anti PD-L1 antibody therapy, chemotherapy, radiotherapy, targeted therapy;
  2. Received any investigational medication within 4 weeks prior to the first use of the investigational medication;
  3. Subjects who require systemic treatment with corticosteroids (>10 mg prednisone equivalent dose per day) or other immunosuppressants within 2 weeks prior to the first use of the study drug are excluded from the use of corticosteroids for local esophageal inflammation and prevention of allergies, nausea, and vomiting. Other special circumstances require communication with the sponsor. In the absence of active autoimmune diseases, it is allowed to inhale or locally use steroids and adrenal cortex hormone replacement with a dose greater than 10mg/day of prednisone efficacy dose;
  4. Individuals who have received anti-tumor vaccines or have received live vaccines within 4 weeks prior to the first administration of the investigational drug; 8. Have any history of active autoimmune diseases or autoimmune diseases (such as interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary inflammation, vasculitis, myocarditis, nephritis, hyperthyroidism, hypothyroidism); Excluding patients with vitiligo or those who have recovered from asthma/allergies of the same age and do not require any intervention in adulthood; Patients with autoimmune mediated hypothyroidism treated with thyroid replacement hormone at a stable dose and type I diabetes patients treated with insulin at a stable dose can be included; 9. Have a history of immunodeficiency, including HIV testing positive, or other acquired or congenital immunodeficiency diseases, or a history of organ transplantation and allogeneic bone marrow transplantation; 10. Subjects with uncontrolled clinical symptoms or diseases of the heart, such as (1) NYHA II and above heart failure, (2) unstable angina, (3) myocardial infarction within 1 year, and (4) clinically significant supraventricular or ventricular arrhythmias requiring clinical intervention; 11. Serious infections (CTC AE>Level 2) occurred within 4 weeks prior to the first use of the investigational drug, such as severe pneumonia, bacteremia, and infection complications that require hospitalization treatment; Baseline chest imaging examination suggests the presence of active pulmonary inflammation and symptoms and signs of infection within 2 weeks prior to the first use of the study drug, requiring oral or intravenous antibiotic treatment, except for prophylactic antibiotic use; 12. Have a history of interstitial lung disease and non infectious pneumonia, and pulmonary function tests confirm ≥ grade 3 pulmonary insufficiency; 13. Patients who have been diagnosed with active pulmonary tuberculosis infection through medical history or CT examination, or have a history of active pulmonary tuberculosis infection within one year before enrollment, or have a history of active pulmonary tuberculosis infection more than one year before but have not received formal treatment; 14. The subject has active hepatitis B (HBV DNA ≥ 2000 IU/mL or 104 copies/mL), hepatitis C (hepatitis C antibody positive, and HCV RNA above the detection limit of the analysis method); 15. There are abnormal laboratory test values of sodium, potassium, and calcium greater than level 1 within the first two weeks of enrollment, which cannot be improved after treatment; 16. Known allergic reactions, hypersensitivity reactions, or contraindications to macromolecular protein preparations, or any components of serplulimab, or to paclitaxel or cisplatin or any components used in their preparations; 17. Diagnosed as any other malignant tumor before the first use of the investigational drug, excluding malignant tumors with low risk of metastasis and death (5-year survival rate>90%), such as basal cell or squamous cell skin cancer or cervical cancer in situ that has been adequately treated; 18. According to the judgment of the researchers, the subjects may have other factors that may force them to terminate the study midway, such as having other serious illnesses (including mental illness) that require concurrent treatment, having other serious illnesses (such as myocardial infarction, cerebrovascular accident) in the near future, high risk of recurrence, severe abnormalities in laboratory test values, family or social factors, which may affect the safety of the subjects or the collection of trial data.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
mPFS | up to one year
  Median Progression-Free-Survival

SECONDARY OUTCOMES:
ORR | through study completion, an average of 18 month
  overall response rate
OS | through study completion, an average of 18 month
  Overall Survival
DOR | through study completion, an average of 18 month
  During of response
Toxic side reactions | through study completion, an average of 18 month
  The US Toxicity Evaluation Standard (CTC5.0) is divided into O~4 grades, and the evaluation of acute radiation reactions adopts RTOG/EROTC criteria

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No